CLINICAL TRIAL: NCT05475925
Title: A Multicenter, Open-Label, First-In-Human, Multiple Expansion Cohort, Phase 1/2 Study to Evaluate the Safety and Efficacy of DR-01 in Adult Subjects With Large Granular Lymphocytic Leukemia or Cytotoxic Lymphomas
Brief Title: A Study of DR-01 in Subjects With Large Granular Lymphocytic Leukemia or Cytotoxic Lymphomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dren Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DR-01-ONC-001
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: LGLL - Large Granular Lymphocytic Leukemia; Primary Cutaneous Gamma-Delta T-Cell Lymphoma; Primary Cutaneous CD8+ Aggressive Epidermotropic T-Cell Lymphoma; Hepatosplenic T-cell Lymphoma; Subcutaneous Panniculitis-Like T-Cell Lymphoma; Aggressive NK Cell Leukemia; Systemic EBV1 T-cell Lymphoma, if CD8 Positive; Hydroa Vacciniforme-Like Lymphoproliferative Disorder; Extranodal NK/T Cell Lymphoma, Nasal Type; Enteropathy-Associated T-Cell Lymphoma; Monomorphic Epitheliotropic Intestinal T-Cell Lymphoma; Cytotoxic PTCL-NOS (CD8+ or CD56+ and Cytotoxic Marker); Cutaneous PTCL-NOS (CD8+ or CD56+ and Cytotoxic Marker)
Keywords: LGLL; Cytotoxic; Lymphoma; ANKL; EATL; MEITL; ENKL; HSTCL; Leukemia; SPTCL; ENKTL; CTCL; PTCL-NOS; TCL
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Subcutaneous panniculitis-like T-cell lymphoma; Lymphoma, Extranodal NK-T-Cell; Enteropathy-Associated T-Cell Lymphoma; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A Dose Escalation 1 mg/kg of DR-01 (Experimental): Subjects in this arm will initially receive 1 mg/kg at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing (up to 6 mg/kg) thereafter for up to 25 cycles total.
  Interventions: Drug: DR-01
- Part A Dose Escalation 3 mg/kg of DR-01 (Experimental): Subjects in this arm will initially receive 3 mg/kg at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing (up to 10 mg/kg) thereafter for up to 25 cycles total.
  Interventions: Drug: DR-01
- Part A Dose Escalation 6 mg/kg of DR-01 (Experimental): Subjects in this arm will initially receive 6 mg/kg at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing (up to 10 mg/kg) thereafter for up to 25 cycles total.
  Interventions: Drug: DR-01
- Part A Dose Escalation 10 mg/kg of DR-01 (Experimental): Subjects in this arm will initially receive 10 mg/kg at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing (up to 10 mg/kg) thereafter for up to 25 cycles total.
  Interventions: Drug: DR-01
- Part A Dose De-escalation 0.3 to <1 mg/kg of DR-01 (Experimental): This cohort would only be triggered should a DLT occur at Dose Level 1 or if recommended by the Safety Review Committee. Subjects in this arm would initially receive 0.3 to <1 mg/kg at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing (up to 3 mg/kg) thereafter for up to 25 cycles total.
  Interventions: Drug: DR-01
- Part B Dose Expansion (Cohort B1) Optimized Dose/Regimen of DR-01 (Experimental): Subjects in this arm will receive the pharmacologically optimized dose/regimen for LGL leukemia subjects determined in Part A. Depending on the selected dose/regimen, subjects will receive target dose at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing thereafter for up to 25 doses total.
  Interventions: Drug: DR-01
- Part B Dose Expansion (Cohort B2) Optimized Dose/Regimen of DR-01 (Experimental): Subjects in this arm will receive the pharmacologically optimized dose/regimen for cytotoxic lymphoma subjects determined in Part A. Depending on the selected dose/regimen, subjects will receive target dose at either the Primary regimen (bi-weekly dosing for fist month), Secondary regimen (doses at Days 1, 8, 15, 29 during first month), or Tertiary regimen (dosing days 1-5, 15, 29 during first month), followed by monthly dosing thereafter for up to 25 doses total.
  Interventions: Drug: DR-01

INTERVENTIONS:
Drug: DR-01 — DR-01 is a non-fucosylated, human immunoglobulin G1 (IgG1) monoclonal antibody.

SUMMARY:
This is a multicenter, first-in-human, Phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and anti-tumor activity of DR-01 in adult patients with large granular lymphocytic leukemia or cytotoxic lymphomas

ELIGIBILITY:
Inclusion Criteria (All Subjects):

1. ≥18 years of age.
2. Able to understand and comply with protocol-required study procedures and voluntarily sign a written informed consent document.
3. Sufficient key organ performance and coagulation.
4. Female subjects of childbearing potential (postmenarcheal, has an intact uterus and at least one ovary, and is <1 year postmenopausal) must agree to use a highly effective method of contraception from enrollment through at least 12 months after last dose of DR-01.
5. Male subjects must agree to use acceptable effective method(s) of contraception.

   Subjects with LGLL must also meet inclusion criteria 6 and 7.
6. Must have discontinued at least one prior line of systemic therapy.
7. Additional immunophenotypic criteria must be met.

   Disease-specific Inclusion Criteria (Cytotoxic Lymphomas):

   Subjects with cytotoxic lymphomas must also meet inclusion criteria 8,9, and 10.
8. Subjects must have failed at least two prior systemic regimens.
9. Availability of post-progression tissue sample or willingness to consent to a baseline biopsy.
10. Histologically confirmed diagnosis of a cytotoxic lymphoma by a hematopathologist (according to the WHO 2016 classification [Swerdlow 2016]).
11. For Part A only, evaluable disease is acceptable.
12. For Part B2 only:

Subjects must have radiographically measurable disease to be assessed by Lugano criteria. Subjects with primary cutaneous variants must have at least 1 measurable lesion that is evaluable using the Olsen criteria (Olsen 2021) or leukemic involvement that can be evaluated using a modified TPLL response criteria (Staber 2019).

Subjects with hepatosplenic disease or other variants that do not have measurable disease by Lugano criteria (Cheson 2014) may be eligible upon discussion with the Medical Monitor if they have identifiable leukemic involvement in BM or peripheral blood (meeting the CD8+ cytotoxic phenotype definition) that can be evaluated for response using a modified TPLL response criteria (Staber 2019), or skin involvement that can be evaluated using Olsen criteria (Olsen 2021).

Exclusion Criteria:

Disease-specific Exclusion Criteria; LGLL and ANKL:

1. A reactive LGL lymphocytosis to a viral infection or LGL associated with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

   The following exclusion criteria apply to all subjects:
2. Active systemic infection or severe localized infection requiring systemic antibiotics, antivirals or antifungals.
3. Active or suspected malignant central nervous system involvement.
4. Life-threatening, severe complications of malignancy (e.g., uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation).
5. Active known second malignancy.
6. Infection with human immunodeficiency virus (HIV) type 1 or 2 (HIV-1 or HIV-2).
7. Hepatitis B infection (hepatitis B virus surface antigen [HBsAg] positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Subjects with HCV with undetectable virus after treatment are eligible.
8. History of clinically significant cardiac disease or congestive heart failure greater than New York Heart Association (NYHA) Class II.
9. Use of systemic corticosteroids (e.g., >5 mg/day prednisone or equivalent for subjects with LGL leukemia (subjects on 20 mg prednisone or equivalent to treat LGL leukemia must be weaned within 28 days post C1D1 to 5 mg) and >10 mg/day prednisone or equivalent for subjects with cytotoxic lymphoma) within 15 days (except for prophylaxis for radiodiagnostic contrast reactions), or other non-biological immunosuppressive drugs within 15 days, prior to C1D1. Patients on stable prednisone ≤10 mg for documented rheumatologic/autoimmune conditions are exempted from this requirement.
10. Any condition requiring hormonal therapy (except for contraception, hormone replacement therapy and hormonal prophylaxis for a prior malignancy).
11. Any other medical or psychiatric condition, or laboratory abnormality that would increase the risk associated with study participation, in the opinion of the Investigator or Medical Monitor.
12. Toxicities from previous anticancer therapies must have resolved to baseline levels or to Grade 1 (except for alopecia, peripheral neuropathy, or hematologic parameters meeting inclusion criteria).
13. Autologous HSCT within 40 days of C1D1, allogeneic HSCT within 90 days
14. Any immunosuppressive therapy for GVHD for subjects who are post allogeneic HSCT.
15. Major surgery within 28 days of C1D1 (requires more than local anesthesia or plexus blockade).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability. To determine the incidence and severity of adverse events as assessed by CTCAE v5.0. | Up to 25 months
Part A: Safety and Tolerability. To determine the incidence and severity of dose limiting toxicities (DLTs) as defined by protocol specified DLT criteria. | During First 28 days (Cycle 1)
Part A: To determine potential pharmacologically optimized dose/regimen for DR-01 in LGL leukemia and cytotoxic lymphoma populations as determined using an integrated assessment of efficacy, safety, PK/PD, and exposure-response relationships. | Up to 6 months
Part B: Overall Response Rate (ORR), defined as the proportion of subjects with Complete Response (CR) or Partial Response (PR) based on disease-specific response criteria. | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Jen Hong, MD, Study Director — Dren Bio
Locations (36):
- United States (14):
  - Dren Investigational Site, Birmingham, Alabama
  - Dren Investigational Site, Duarte, California
  - Dren Investigational Site, Redwood City, California
  - Dren Investigational Site, New Haven, Connecticut
  - Dren Investigational Site, Tampa, Florida
  - Dren Investigational Site, Boston, Massachusetts
  - Dren Investigational Site 1, New York, New York
  - Dren Investigational Site 2, New York, New York
  - Dren Investigational Site, Columbus, Ohio
  - Dren Investigational Site 2, Pittsburgh, Pennsylvania
  - Dren Investigational Site, Houston, Texas
  - Dren Investigational Site, Charlottesville, Virginia
  - Dren Investigational Site, Fairfax, Virginia
  - Dren Investigational Site, Seattle, Washington
- Australia (3):
  - Dren Investigational Site, Clayton, Victoria
  - Dren Investigational Site, Richmond, Victoria
  - Dren Investigational Site, Nedlands, Western Australia
- France (3):
  - Dren Investigational Site, Pierre-Bénite
  - Dren Investigational Site, Rennes
  - Dren Investigational Site, Toulouse
- Germany (3):
  - Dren Investigational Site, Berlin
  - Dren Investigational Site, Cologne
  - Dren Investigational Site, Leipzig
- Hong Kong (2):
  - Dren Investigational Site 1, Hong Kong
  - Dren Investigational Site 2, Hong Kong
- Dren Investigational Site, Bologna, Italy
- South Korea (6):
  - Dren Investigational Site 1, Busan
  - Dren Investigational Site 2, Busan
  - Dren Investigational Site, Goyang-si
  - Dren Investigational Site 1, Seoul
  - Dren Investigational Site 2, Seoul
  - Dren Investigational Site 3, Seoul
- Spain (2):
  - Dren Investigational Site, Barcelona
  - Dren Investigational Site, Salamanca
- Taiwan (2):
  - Dren Investigational Site, Tainan
  - Dren Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: No